

Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

## VE-CIP2001/2021

Velusetrag for the treatment of Chronic Intestinal Pseudo-Obstruction (CIPO). A multicenter, double-blind, placebo-controlled, cross-over, multiple (n=1) trial

| Author: | |
|------------------|-------------------|
| Document status: | Final version 2.0 |
| Release date: | 10-MAY-2023 |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### **Document History**

| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|---|---|---|---|
| Draft<br>Version 0.1 | 04-FEB-2022 | N.A. | N.A. |
| Draft<br>Version 0.2 | 15-FEB-2022 | Internal Review | Internal Review |
| Draft<br>Version 0.3 | 24-MAR-2022 | The following section are updated: 1.1 (to explain why CMH test is not reported); 3.1, 3.3.1, 4.2, 5, 6.2 (minor changes); 6.3.1, 6.3.2 (put reference and further details are included); 6.3.4 (minor changes); 6.4.3, 6.4.4, 6.4.5, 6.4.6 (the baseline used for changes computation is updated); 6.5 (details for subgroup analysis are included) and 8 (appendix of scoring method reported). | Sponsor's review |
| Draft<br>Version 0.4 | 12-APR-2022 | Sections 1.1, 4.4.1, 6.3.2.1 are updated. Minor changes in sections 4.2, 5, 6.3.1, 6.3.2.3, 6.3.2.7, 6.3.2.8, 6.3.2.14, 6.4.5, 6.4.6, 6.5. Description of switch added in section 6.1. | Sponsor's review Internal review |
| Draft<br>Version 0.5 | 30-MAY-2022 | Sections related to efficacy endpoint are updated. | Sponsor's review |
| Draft<br>Version 0.6 | 15-FEB-2023 | Section 1.1 Changes from The Study Protocol, Definition of baseline and first/last administration of study treatment in section 4.2 Definition, section 4.4.2. Handling of Missing Data/Imputation/Censoring Rules, section 6.1 Study subjects, section 6.3.2.6 , section 6.3.2.8 , section | Sponsor's and internal review |



| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|---|---|---|---|
| | | 6.3.2.14. Concentration of velusetrag and THRX-830449 metabolite, section 6.4.4 laboratory parameters and section 6.4.6 other safety parameters are updated. | |
| | | Minor changes are applied for Sections related to efficacy endpoint. | |
| | | "Patient" replaced with "Subject". | |
| | | Start of treatment replaced with pre-<br>treatment. | |
| | | Column "Endpoints" of section 2 updated for safety and tolerability secondary objective. | |
| | | Section 3.3.3 updated included further details to identify prohibited medication. | |
| | | Definition of study phases, Figure 2 and definition of baseline/reference are updated in section 4.2. | |
| | | NOPD03 is included in Table 6.1-1. | |
| Draft<br>Version 0.7 | 13-MAR-2023 | Details related to the sort of outputs of medical history and prior medication are included in section 6.2. The "abnormal" category of physical examination is splitted in "abnormal CS" and "abnormal NCS" in section 6.2. | Sponsor's review |
| | | A listing of and gastrointestinal symptoms is added in section 6.3.1. | |
| | | Descriptive tables by treatment sequence and period are deleted for primary endpoint (section 6.3.1), | |



| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|-----------------------|--------------|--------------------|----------------|



| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|---|---|---|---|
| Final Version<br>1.0 | 15-MAR-2023 | First Final Release | Sponsor's approval |
| | | Section 1.1 is updated to report the decision to not considered the variable stratum in the efficacy analyses and all efficacy sections are updated consequently (i.e., 6.3.1, 6.3.2.1, 6.3.2.2, 6.3.2.4, 6.3.2.8). Section 6.1 is updated to better clarify how subject disposition will be described | |
| Draft<br>Version 1.1 | 20-APR-2023 | and to drop tables by stratum. Time from CIPO diagnosis date to informed consent signature described in Section 6.2 is computed in years instead of months. | Sponsor's review |
| | | The analysis of primary endpoint on FAS is removed in section 6.3.1. | |
| | | Section 6.3.2.9 related to is updated including additional details. | |
| | | Section 6.3.2.11 and section 6.3.2.13 are updated to consider the variables as | |



| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|---|---|---|---|
| | | categorical and to include data collected for wash-out/follow-up period and statistical model for are removed. | |
| | | Formal adjustment for section 6.4.3. | |
| | | Further details are included for listings with abnormal values in section 6.4.4 and 6.4.6. | |
| | | are updated in section 6.4.4. | |
| | | Section 1.1 updated with further details on binary outcome and count data. Fisher exact test was included in the section 6.3.2.2 and 6.3.2.13. | |
| | | ATC codes to identify opioids treatments is section 3.3.3 were update as well as the ATC code to identify patients who took antibiotics in section 6.3.2.7. | |
| Draft<br>Version 1.2 | 09-MAY-2023 | Including also start date for prior medications (including the start date of medical history condition on which imputation rules for partial dates will be applied to compute the study day. | Sponsor's review |
| | | Management of collected with different unit of measurements where there isn't conversion faction applicable to uniform the unit are described for | |
| | | Similarly, management of collected as greater than (>) or lower than (<) will be also described. | |
| | | Mixed models for efficacy parameters considered as continuous variables were updated considering the reference of | |



| Status and<br>Version | Release Date | Change Description | Reason/Comment |
|---|---|---|---|
| | | Model 2 described in the publication of Chen X, Chen P "A Comparison of Four Methods for the Analysis of N-of-1 Trials" PLoS One. 2014 Feb 4;9(2):e87752. doi: 10.1371/journal.pone.0087752. eCollection 2014. Due to the different approach adopted for continuous variables, the Mixed model planned for binary outcome was removed also due to possible convergence problems. | |
| | | The McNemar Bowker's test planned for and was replaced with Fisher exact test to compare treatment. Formal adjustments. | |
| Final Version<br>2.0 | 10-MAY-2023 | Second Final Release | Sponsor's approval |



### Authorization

The signatures on this page indicate review and approval of the Statistical Analysis Plan, version 2.0, dated May 10, 2023.

| | Name | Function | Signature | Date |
|---|---|---|---|---|
| Author | | | DocuSigned by: Signer Name: Signing Reason: I am the au Signing Time: 10-May-2023 | thor of this documen<br>18:41 CEST |
| Reviewer | | | DocuSigned by: Signer Name: Signing Reason: I have revising Time: 10-May-2023 | ewed this document<br>18:46 CEST |
| Alfasigma S.p.A | | | DocuSigned by: Signer Name: Signing Reason: I approve the Signing Time: 10-May-2023 | is document<br>19:31 CEST |
| Alfasigma S.p.A | | | DocuSigned by: Signer Name: Signing Reason: I approve to Signing Time: 10-May-2023 | his document<br>23:00 CEST |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### **TABLE OF CONTENTS**

| LIST OI | ABBRE | VIATIONS | 11 |
|---|---|---|---|
| 1. | INTRO | DUCTION | 13 |
| 1.1. | CHANGES FROM THE STUDY PROTOCOL | | |
| 2. | STUDY | OBJECTIVES AND ENDPOINTS | 14 |
| 3. | ВАСКО | GROUND AND RATIONALE | 19 |
| 3.1. | OVERA | ALL STUDY DESIGN AND PLAN DESCRIPTION | 19 |
| 3.2. | SELECT | FION OF STUDY POPULATION | 21 |
| 3.3. | TREAT | MENT | 22 |
| | 3.3.1. | Treatment Administered | 22 |
| | 3.3.2. | Method of Assigning Subjects to Treatment Group | 22 |
| | 3.3.3. | Prior and Concomitant Therapy | 23 |
| 3.4. | SCHED | ULE OF TIME AND EVENTS | 26 |
| 3.5. | SAMPL | LE SIZE AND POWER ESTIMATION | 29 |
| 4. | DEFIN | ITIONS AND GENERAL METHODOLOGY | 30 |
| 4.1. | .1. GENERAL METHODOLOGY | | 30 |
| 4.2. | DEFINI | ITIONS | 30 |
| 4.3. | CODIN | IG OF THERAPIES AND MEDICAL TERMS | 32 |
| 4.4. | HANDI | LING OF DROP-OUTS OR MISSING DATA | 33 |
| | 4.4.1. | Missing or Partial Dates | 33 |
| | 4.4.2. | Handling of Missing Data/Imputation/Censoring Rules | 33 |
| | 4.4.3. | Handling of Drop-Out Subjects | 34 |
| 4.5. | MULTI | PLE COMPARISON/MULTIPLICITY | 34 |
| 4.6. | MULTI | CENTRE STUDIES/CENTER POOLING | 34 |
| 5. | ANALYSIS POPULATIONS | | |
| 6. STATISTICAL METHODOLOGY | | STICAL METHODOLOGY | 35 |
| 6.1. | STUDY | SUBJECTS | 35 |
| 6.2. | BACKG | GROUND AND DEMOGRAPHIC CHARACTERISTICS | 37 |
| 6.3. | EFFICA | CY EVALUATION | 39 |
| | 6.3.1. | Primary efficacy analysis | 39 |
| | 6.3.2. | | 41 |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



6.4.

| 8. | | APPENDIX | 59 |
|----|------|--------------------------------------|----|
| 7. | | REFERENCES | 59 |
| | 6.6. | INTERIM ANALYSIS AND DATA MONITORING | 59 |
| | 6.5. | SUBGROUP ANALYSES | 59 |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### **LIST OF ABBREVIATIONS**

5-HT<sub>4</sub> 5-hydroxytryptamine receptor 4

AE Adverse event

ALP Alkaline phosphatase

ALT Alanine aminotransaminase

API Active pharmaceutical ingredient

AST Aspartate aminotransferase

ATC Anatomical Therapeutic Chemical

BMI Body mass index

BP Blood pressure

CH<sub>4</sub> Methane

CIPO Chronic intestinal pseudo-obstruction

CRF Case report form

CSR Clinical Study Report

CYP(3A4) Cytochrome P450 (isozyme 3A4)

ECG Electrocardiogram

eCRF Electronic-case report form

EFU End of follow up

EOT End of treatment

ES Effect size

ESV Early switch visit

ETV Early termination visit

FAS Full analysis set



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

H<sub>2</sub> Hydrogen

ICF Informed consent form

IWRS Interactive web response system

LOCF Last observation carried forward

MedDRA Medical Dictionary for Regulatory Activities (MEDDRA®)

mFAS Modified full analysis set

NOPD Non-protocol deviation

PPS Per protocol set

PT Preferred term

\_\_\_\_

SOC System organ class

SOT Start of treatment

SS Safety set

T3 Triiodothyronine

T4 Thyroxine

\_\_\_\_

TSH Thyroid stimulating hormone

ULN Upper Limit of Normal

WHO-DD World Health Organization Drug Dictionary



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### 1. INTRODUCTION

This statistical analysis plan (SAP) provides details on the planned statistical analysis for study VE-CIP2001/2021 (CIPO) based on the study protocol final version 1.0 of May 24, 2021.

### 1.1. Changes from The Study Protocol

| The endpoints " | |
|---|---|
| " reported in section 5.2 SECONDARY | STUDY OBJECTIVES AND ENDPOINTS o |
| study protocol are analysed | |
| The Handling of Missing and Incomplete Data for | primary endpoint has been modified in |
| case of pre-treatment value missing. | |
| The reason for this is to reduce data heterogenei | ty between subjects |

In addition, missing imputation methodology will be applied only for the primary endpoint of the study while all other secondary endpoints will be based on observed data. For this reason, the rules explained in section 16.3.5 Handling of Missing and Incomplete Data of study protocol for the other endpoints are not reported since not applied.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

Number of and number of will be analyzed as categorical variables and will be separately analyzed for treatment and washout/follow-up period.

### 2. STUDY OBJECTIVES AND ENDPOINTS

| OBJECTIVES | VARIABLES | ENDPOINTS |
|---|---|---|
| Primary study objective: | | Primary study endpoint: |
| To investigate the efficacy of velusetrag in improving the symptoms severity associated with CIPO, in subjects with idiopathic CIPO and CIPO | Rating of each symptom (i.e., abdominal pain, bloating, nausea and vomiting) using a Likert scale from 0=Absent to 4= | Change in weekly global gastrointestinal symptoms average index score* from pretreatment to the end of each treatment period. |
| secondary to neurodegenerative or demyelinating conditions (e.g., Parkinsonian Syndromes, multiple sclerosis etc.). | Extremely severe (precluding daily activities). | *The weekly global gastrointestinal symptoms average index score is obtained by averaging the scores for each of the 4 symptoms assessed weekly: abdominal pain, bloating, nausea and vomiting. |
| | | Rating of symptoms (i.e. abdominal pain, bloating, nausea and vomiting) is using a recall period of 7 days and a Likert scale with the following categories: |
| | | 0 – Absent |
| | | 1 - Mild (not influencing usual activities) |
| | | 2 - Moderate (diverting from, but not urging modification of, usual activities) |
| | | 3 - Severe (influencing usual activities markedly enough to urge modifications) |



| OBJECTIVES | VARIABLES | ENDPOINTS |
|------------|-----------|----------------------------------------------------|
| | | 4 - Extremely severe (precluding daily activities) |



| OBJECTIVES | VARIABLES | ENDPOINTS |
|------------|-----------|-----------|



| OBJECTIVES | VARIABLES | ENDPOINTS |
|------------|-----------|-----------|



| OBJECTIVES | VARIABLES | ENDPOINTS |
|------------|-----------|-----------|
| | | - |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



### 3. BACKGROUND AND RATIONALE

### 3.1. Overall Study Design and Plan Description

This is a phase II, multicenter, double-blind, placebo-controlled, two-treatment four-period cross-over, multiple (n=1) trial to evaluate the efficacy and safety of velusetrag 15 mg once a day, compared to placebo, in subjects with a diagnosis of idiopathic CIPO or CIPO secondary to primary neurodegenerative or demyelinating conditions (e.g., Parkinsonian Syndromes, multiple sclerosis, etc.).

Eligible subjects will be treated for 4 periods of 4 weeks each with either velusetrag 15 mg (2 periods) or placebo (2 periods), once daily, with a wash-out period of 2 weeks between treatment periods. The scheme of study design is provided in Figure 1 below.

Figure 1: Schematic study design



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



After an up to 7-day screening period (from Day -7 to Day -1, V1), at randomization visit (V2), eligible subjects will be randomly allocated to one of the following four sequences:

A. VEL-PLA-VEL-PLA

B. PLA-VEL-PLA-VEL

C. VEL-PLA-PLA-VEL

D. PLA-VEL-VEL-PLA

#### Where:

VEL= velusetrag 15 mg once daily for 4 weeks.

PLA= matching placebo once daily for 4 weeks.

There will be a 2-week wash-out period between each treatment period and a final 2-week follow-up period at the end of the last treatment period.

Subjects will be assessed during a total of 10 visits during the study, as detailed in the Study Schedule of Assessments, including the screening visit, a start of treatment visit (SOT) and an end of treatment visit (EOT) for each of the 4 treatment periods, for a total of 8 visits, and a final End of Follow up Visit (EFU), 2 weeks after the end of the last treatment period.

If the subject cannot go back to the clinical center for one or more of the following visits: EOT- 2 (Visit 5), EOT- 3 (Visit 7), EOT- 4 (Visit 9), End Of Follow Up (EFU, Visit 10) or in case of an early termination visit (ETV), the visit will be scheduled at the subject's home and will be performed by a home nursing service. The clinical study staff at the clinical center may also attend the visit remotely.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

Overall, each subject will be involved in the study for a screening period of up to 7 days before randomization and approximately a 24-week period after randomization.

Subjects under treatment with a must have a 5-day wash-out period before randomization (note: symptomatic treatments other than see section 10.8 Prior and Concomitant Therapy in the study protocol).

If, during a treatment period or during a wash-out period, a subject should experience an exacerbation of CIPO related gastrointestinal symptoms that is not controlled by permitted medications and is not judged as an adverse event, he/she will attend an early switch visit (ESV) at the clinical site. After being reassessed, he/she will be offered to directly switch to the next scheduled treatment period (SOT-2 or SOT-3 or SOT-4) without completing the ongoing treatment or wash-out period. Only one early switch is possible during the study. ESV will be Day 1 of the relevant period (SOT-2 or SOT-3 or SOT-4) based on the timing of early switch.

In case of ESV/SOT-2 or ESV/SOT-3 or ESV/SOT-4, the subsequent visits will follow the relevant sequential number (see Study Schedule of Assessments in section 3.4).

### 3.2. Selection of Study Population

Sixteen male and female subjects with a diagnosis of idiopathic CIPO or CIPO secondary to primary neurodegenerative or demyelinating conditions (e.g., Parkinsonian Syndromes, multiple sclerosis, etc.) who meet all the inclusion and none of the exclusion criteria will be enrolled in this study.



Subjects will be enrolled in up to 5 centres.

A complete list of all inclusion criteria and exclusion criteria are provided in Section 9.2 and 9.3 of the study protocol, respectively.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

#### 3.3. Treatment

#### 3.3.1. Treatment Administered

The investigational products that will be administered in the study were:



### 3.3.2. Method of Assigning Subjects to Treatment Group

Eligible subjects will be randomly allocated in a 1:1:1:1 manner (4 subjects per treatment sequence), in a blinded fashion, to one of the following four treatment sequences:

- A. VEL-PLA-VEL-PLA
- B. PLA-VEL-PLA-VEL
- C. VEL-PLA-PLA-VEL
- D. PLA-VEL-VEL-PLA

#### Where:

VEL= velusetrag 15 mg ( mg once a day for 4 weeks. PLA= matching placebo ( ) once a day for 4 weeks.

Since the study is a cross-over study, each subject will take both investigational products during the study according to treatment sequence assigned by randomization.

Randomization will be stratified into 3 strata by CIPO diagnosis (idiopathic or secondary to neurodegenerative or demyelinating disease) and by responder status (responder/naive or non-responder) as follows:

non-responderresponder/naïve and idiopathic CIPO



Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

• responder/naïve and CIPO secondary to neurodegenerative or demyelinating disease.

Non responders are defined as all subjects that, based on investigator's judgement, have an history of a lack of benefit

### 3.3.3. Prior and Concomitant Therapy

Use of the following <u>medications is not allowed</u> within 2 weeks prior to Screening and/or planned throughout the duration of the study:

- Scopolamine
- Erythromycin
- Strong CYP3A4 inhibitors or strong CYP3A4 inducers.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

| (not exhaustive list*) |
|------------------------|

• Strong P-gp transporter inhibitors.

| Strong P-gp | Inhibitors |
|-------------|------------------------|
| | (not exhaustive list*) |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

• Strong BCRP transporter inhibitors.

In addition, use of:

- Opioids is not allowed within 8 weeks from screening and/or planned throughout the duration of the study.
- are not allowed starting from 5 days before randomization and throughout the duration of the study

Orally poorly absorbed opioids that could be used to treat potential adverse events, such as diarrhea, may be used if medically indicated.

If a or scopolamine, or erythromycin and an opioid for analgesic use is taken during the study, the subject will be considered a treatment failure and will be withdrawn from the study.

Additional prescription and over-the-counter <u>medications are permitted</u>, provided that such agents are not known to be strong inducers or inhibitors of CYP3A4, P-gp and BCRP activity.

<sup>\*</sup>As the list of prohibited agents is not exhaustive, the selection of prohibited medications done by using ATC and PT will be confirmed through a medical review of all concomitant medications (including medications for CIPO)



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

The selection of prohibited medications will be done by using ATC and PT and it will be reviewed and confirmed through a medical review of all concomitant medications (including medications for CIPO).

Any addition or change in regimen of concomitant medications that affect CYP3A4, P-gp and BCRP activity should be in accordance with inclusion or exclusion criteria and recorded in the source documents and the electronic-case report form (eCRF).

<u>Medication(s)</u> used to relieve main symptoms of CIPO are allowed and the use of the following concomitant medications will be registered in the e-diary daily:

- Treatments for nausea and vomiting and/or non-serotoninergic prokinetics.
- Treatments for constipation.
- Treatments for diarrhea.
- Treatments for abdominal pain.
- Others (e.g., octreotide, somatostatin, pancreatic enzymes, probiotics, rifaximin, metronidazole, fluconazole, etc.).

Further details on prohibited and permitted medications are reported in Section 10.8 PRIOR AND CONCOMITANT THERAPY of the study protocol.

#### 3.4. Schedule of Time and Events

The schedule of assessments is shown in Table 3.4.1.

**Table 3.4.1: STUDY SCHEDULE OF ASSESSMENTS** 

| | рc | | eatment<br>riod <sup>a</sup> | | atment<br>iod <sup>a</sup> | | atment<br>iod <sup>a</sup> | | atment<br>od <sup>a</sup> | EFU <sup>n</sup> | ETV | ESV ° |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Period | Randomiz.<br>SOT-1 | EOT-1 | SOT-2 | EOT-2 | SOT-3 | EOT-3 | SOT-4 | EOT-4 | End of Follow-<br>up | Early<br>Termination<br>Visit | Early switch<br>Visit |
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | ETV | ESV |
| Day | -7 to<br>-1 | 1 | 28(±1) | 43(±1) | 70(±1) | 85 (±1) | 112(±1) | 127(±1) | 154(±1) | 169(±1) | | Any time<br>between<br>Day 1<br>and 126 |
| Informed Consent | Х | | | | | | | | | | | |
| On Site Visit | Х | Х | Х | Х | | Х | | Х | | | | Х |
| On Site Visit or home visit <sup>b</sup> | | | | | Х | | Х | | Х | Х | Х | |
| Medical, surgical history and previous medications | Х | | | | | | | | | | | |



| | ъ | | eatment<br>riod <sup>a</sup> | | atment<br>iod <sup>a</sup> | | atment<br>iod <sup>a</sup> | | atment<br>od <sup>a</sup> | EFU " | ETV | ESV ° |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Period | Randomiz.<br>SOT-1 | EOT-1 | SOT-2 | EOT-2 | SOT-3 | EOT-3 | SOT-4 | EOT-4 | End of Follow-<br>up | Early<br>Termination<br>Visit | Early switch<br>Visit |
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | ETV | ESV |
| Assessment of responder status | х | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | |
| | | I | | | | | I | I | I | | | |
| | | | | I | I | | | | | ı | | I |
| | | | | | | | I | I | | ı | | I |
| | | | | | | | I | | | | | I |
| | | | | ı | | ı | ı | ı | ı | ı | | ı |
| | | | | | | ı | | ı | | ı | | ı |
| - | | | | | | | | | | | | |
| | I | | I | | | | | | | | | |
| | | | I | | | ı | I | | | | | I |
| Inclusion/<br>Exclusion Criteria<br>Evaluation | Х | Х | | | | | | | | | | |
| Randomization | | Х | | | | | | | | | | |
| | | ı | I | ı | I | ı | I | I | I | I | | I |
| | | | | I | | | | | | | | I |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

| | po | | eatment<br>riod <sup>a</sup> | | atment<br>od <sup>a</sup> | | atment<br>iod <sup>a</sup> | | atment<br>iod <sup>a</sup> | EFU " | ETV | ESV º |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening Period | Randomiz.<br>SOT-1 | EOT-1 | SOT-2 | EOT-2 | SOT-3 | EOT-3 | SOT-4 | EOT-4 | End of Follow-<br>up | Early<br>Termination<br>Visit | Early switch<br>Visit |
| Visit | V1 | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | ETV | ESV |
| Drug dispensing | | Х | | Х | | Х | | X | | | | Х |
| Drug administration time recording <sup>k</sup> | | х | Х | Х | Х | X | х | X | х | | | Х |
| Drug accountability | | | Х | | Х | | Х | | Х | | Х | X |

SOT: Start of Treatment; EOT: End of Treatment; EFU: End of Follow up; ETV: Early Termination Visit; ; ESV: Early Switch Visit.

- a. Subjects will undergo a 2-week wash-out period between treatment periods.
- b. If the subject cannot go back to the clinical site for one or more of the following visits: Visit 5, 7, 9 and 10 or ETV, they can be performed at the subject's home.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

- k. Dose to be taken under observation at each scheduled visit at the clinical center. The exact time of dose administration should be recorded at all visits.
- I. If the subject cannot go back to the clinical center for Visit 5, 7, 9 or ETV, the empty packs and the unused investigational product of the relevant period will be collected by the study nurse during the home visit.
- m. In all subjects on V2 and V3, blood samples will be collected time of collection must be recorded for each sample.
- n. The final 2 week follow up period are considered also as final 2 week wash out period for the 4th treatment period.
- o. In case, during a treatment period or during a washout period, a subject should experience an exacerbation of the CIPO related gastrointestinal symptoms that is not controlled by permitted medications and is not judged as an adverse event, he/she will attend an early switch visit (ESV) at the site. After being reassessed, he/she will start the next scheduled treatment period (SOT-2 or SOT-3 or SOT-4), without completing the ongoing treatment or washout period. ESV will be Day 1 of the relevant period (SOT-2 or SOT-3 or SOT-4) based on the timing of early switch. Only one early switch is allowed during the study.

### 3.5. Sample Size and Power Estimation

The sample size is based on the main analysis (t-test) of the primary endpoint, which consists in the differences between velusetrag and placebo within each paired treatment cycle (2 per subject).



With a two-sided significance level of 5%, the planned sample size will lead to power levels above 80% to detect effect size (ES) above 0.7 (see table 3.5.1 below).

Table 3.5.1 Power for different values of effect size and number of pairs

| Power for different values of Effect Size* and number of pairs | | | |
|---|---|---|---|
| Number of pairs | ES: 0.6 | ES: 0.7 | ES: 0.8 |
| 18 | 67% | 80% | 89% |
| 24 | 80% | 91% | 96% |
| 28 | 86% | 94% | 98% |
| 32 | 91% | 97% | 99% |

<sup>\*</sup> More than medium to moderate effect size (Cohen, 1988) Estimates obtained using SAS PROC POWER

If based on a blinded review of the data the rate of missing pairs is found to be higher, the sample size might be increased by the Sponsor.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### 4. DEFINITIONS AND GENERAL METHODOLOGY

### 4.1. General Methodology

Statistical tables, figures, listings and analyses will be produced using SAS® for Windows release 9.4 or later (SAS Institute Inc., Cary, NC, USA).

Data from all sites will be pooled and summarized. Continuous data will be summarized by the number of observations, mean, standard deviation (SD), median, first and third quartiles (i.e., 25<sup>th</sup> and 75<sup>th</sup> percentiles), minimum and maximum. Categorical data will be presented by absolute and relative frequencies (n and %).

All efficacy analyses have the objective to show the superiority of velusetrag over placebo. All statistical analysis will be two-sided at a nominal level of 5%. Confidence intervals will be set at the 95% level.

#### 4.2. Definitions

### Study Phases

**Screening phase (i.e., Visit 1):** the screening phase is defined as starting from the screening visit up to randomization.

The screening visit can be performed within Day -7 and Day -1 before randomization.

**First treatment period** running from Visit 2 to Visit 3 and corresponding to the first period in which subjects took the first treatment assigned at randomization according to treatment sequence.

Wash-out after first treatment period corresponds to the 2-weeks after Visit 3 (EOT-1) in which subjects will not take any investigational product.

Similarly, there will be a **second, third and fourth treatment period** running from each respective start of treatment visit (SOT-2, SOT-3 and SOT-4) to each end of treatment visit (EOT-2, EOT-3 and EOT-4) after 28 days.

Wash-out periods after second and third treatment period corresponds to the 2 weeks after EOT-2 and EOT-3 respectively. Finally, the **follow-up of 2-weeks** corresponds to the 2 weeks after the EOT-4. During these phases the subject will not take any investigational product.

### <u>Definition of cycles</u>

Each subject will be followed for two cycles of both treatments (i.e., VEL-PLA or PLA-VEL). The 1<sup>st</sup> cycle is made up of Period 1 and Period 2. The 2<sup>nd</sup> cycle is made up of Period 3 and



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

Period 4. In the Figure 2 below there are represented period and cycle based on study design.

Figure 2: Schematic design of period and cycle



### **Definition of Screening Failures**

A screening failure is defined as a subject who signs the informed consent and has not been randomized to treatment.

### Definition of Baseline/Reference

Due to the cross-over study design structure, for efficacy evaluation Baseline (for Period 1)/Reference (for Period 2, 3, 4) values are the last values collected prior to each treatment period initiation. For eDiary data the Baseline/Reference values are those recorded at the day before the start of treatment visit (Day -1 for Period 1, end of wash-out for the Period 2, 3, 4), while for other variables recorded in eCRF the Baseline/Reference are the last values collected before each treatment period first intake.

The Baseline for changes computation for the safety assessments is at the Visit 2 (SOT-1) except for laboratory data that is Visit 1.

For efficacy evaluation after the discontinuation of each treatment, the reference for changes computation is defined as the end of treatment visit for each period: Visit 3 (EOT-1) for period 1, Visit 5 (EOT-2) for period 2, Visit 7 (EOT-3) for period 3 and Visit 9 (EOT-4) for period 4.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

In case of early switch visit or premature interruption of treatment, the reference for changes computation within each period should be adjusted accordingly based on ESV visits.

### First/Last Administration of Study Treatment

Considering the overall study, the date of first administration of treatment (i.e., velusetrag or placebo) is the earliest start date of the 4 periods reported in the "Study treatment dispensed" CRF page while the date of last administration of treatment (i.e., velusetrag or placebo) is the date reported in the "End of treatment disposition" CRF page (i.e., maximum of the last administration of the 4 periods).

According to the study design, subjects will not receive the treatment during the wash out periods. For each study period, the date of first administration of treatment is the start date reported in the "Study treatment dispensed" CRF page on the corresponding SOT visit (i.e., Visit 2 (SOT-1) for period 1, Visit 4 (SOT-2) for period 2, Visit 6 (SOT-3) for period 3 and Visit 8 (SOT-4) for period 4)) while the date of last administration of treatment is the last treatment intake date reported in the "Study treatment returned" CRF page on the corresponding EOT visit (i.e., Visit 3 (EOT-1) for period 1, Visit 5 (EOT-2) for period 2, Visit 7 (EOT-3) for period 3 and Visit 9 (EOT-4) for period 4). In case of early switch visit or premature interruption of treatment, the first and last intake within each period should be adjusted accordingly.

#### Study day

The study day describes the day of the event or assessment date relative to the reference start date, which is defined as the date of Randomization.

The study day will be calculated as the difference between the date of each considered efficacy/safety assessment and the reference start date plus 1 day.

If the considered event starts before the Randomization date, the study day will be calculated as the difference between the date of the assessment and the reference start date. Therefore, the study day will be negative.

### 4.3. Coding of Therapies and Medical Terms

The World Health Organization Drug Dictionary (WHO-DD) Version\_B3\_Q1\_2021 will be used to code medications reported in the prior medication, concomitant medication and medications for CIPO (gastrointestinal symptoms) eCRF pages.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

The Medical Dictionary for Regulatory Activities (MedDRA) English version 24.0 will be used to code medical terms reported in the Medical History, non-drug therapies or surgical and medical procedures and Adverse Events eCRF pages.

At the end of the study, if an updated version of the dictionaries is available, dictionaries will be updated after Sponsor's approval, if needed.

### 4.4. Handling of Drop-Outs or Missing Data

### 4.4.1. Missing or Partial Dates

For incomplete dates, the imputation will be performed according to the following rule:

- If the date is completely missing, no imputation will be performed
- In case of day missing, the day will be replaced with 15
- In case of day and month missing, the day will be replaced with 1, the month with July

The imputation rules will be applied to the date of CIPO diagnosis, start date for prior medications (including the condition, start date for concomitant medications (including the medications for CIPO) and adverse events.

In case that these rules led to CIPO diagnosis later than the informed consent date, CIPO diagnosis will be imputed as the informed consent date. Similarly, in case that imputations led to start date later than the end date for concomitant medications and adverse events, the 1<sup>st</sup> day of the month will be imputed instead of the 15<sup>th</sup>.

### 4.4.2. Handling of Missing Data/Imputation/Censoring Rules

The following rules to impute missing data will be applied for the efficacy primary endpoint and further details are provided in section 6.3.1.

Missing pairs (treatment difference velusetrag minus placebo) can occur when at least one of the following is missing:

- Pre-treatment velusetrag value missing
- End of treatment velusetrag value missing
- Pre-treatment placebo value missing
- End of treatment placebo value missing





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

These rules of imputation will be applied only if a subject starts the period of interest (i.e., if he/she performs the corresponding start of treatment visit).

The above approach will be used for the FAS and as sensitivity analysis for mFAS1, PPS.

No missing imputation will be applied for secondary efficacy endpoints.

### 4.4.3. Handling of Drop-Out Subjects

Subjects who discontinue the study for any reason will be analyzed for efficacy and safety purposes.

### 4.5. Multiple Comparison/Multiplicity

Not applicable.

### 4.6. Multicentre Studies/Center Pooling

The data from all sites will be pooled and analyzed. Given the small sample size, no analysis will be performed by site or country.

### 5. ANALYSIS POPULATIONS

The following analysis populations are defined based on the study protocol:

- Screened population: all subjects who provided informed consent. A screening failure is defined as a screened subject who has not been randomized to treatment.
- Randomized population: all screened subject who has been randomized to treatment.
- Safety Set (SS): all treated subjects (i.e., subject who received at least one
  investigational product or placebo).
- Full Analysis Set (FAS): all randomized and treated subjects.
- Modified Full Analysis Set 1 (mFAS1): all subjects responder/naïve to
   randomized and treated who reported data on the primary endpoint at least
   once during a velusetrag treatment period and at least once during a placebo treatment
   period in the same cycle.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

• **Per Protocol Set (PPS):** all subjects in the mFAS1 who fulfil the study protocol requirements in terms of compliance to treatment and collection of primary efficacy data, and with no major deviations that may affect study results.

For the PPS analysis, if within a period, the compliance is below 80%, the primary endpoint data of this period will be excluded from the analysis. E.g., if compliance data are 100%, 100%, 60%, 60%, the subject is included in the PPS (overall compliance at 80%) but the observations of the third and fourth period are excluded.

The complete list of deviations will be defined in a specific protocol deviation handling plan and a blind data review meeting will occur prior to unblinding. The decisions for exclusion of subjects from the PPS will be taken in a blinded manner and documented.

Analysis on the SS will be performed according to the actual treatment received.

The number of subjects who complete the screening phase

Analysis on the FAS, mFAS1, will be performed according to the treatment and stratum assigned at randomization following the intent-to-treat principle.

Analysis on the PPS will be performed according to the actual stratum, while no cases of study treatment different from the randomized one can belong to the PPS (i.e., subjects receiving a study treatment different from the randomized one will be excluded from the PPS).

### 6. STATISTICAL METHODOLOGY

### 6.1. Study Subjects

| | and the number of subjects who discontinue the |
|---|---|
| screening phase | |
| . , | eason for discontinuation will be summarized overall on per of randomized subjects included will also be displayed. |
| Subject disposition will be provide | d on the randomized population by treatment sequence |
| and overall summarizing the num | ber of subjects randomized and the number of treated |
| subjects. The number of subject | ts who complete the treatment |
| | and the number of subjects |
| who discontinue the treatment | |
| | together with the reason for study discontinuation will |
| be provided. Similarly, the number | of subjects who complete the study |
| | and the number of subjects who |



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

discontinue the study together with the reason for study discontinuation will be provided.

In addition, the number of subjects who enter in each period including wash-out/follow-up (i.e., performed the corresponding SOT visit) and the number of subjects who complete the treatment, who perform switch in treatment period, who discontinue the treatment together with the reason for treatment discontinuation, who complete wash-out/follow-up, who perform switch in the wash-out period or who discontinue the wash-out/follow-up will be also provided considering each period.



The numerousness of the analysis populations (SS, FAS, mFAS1, and PPS) will be described and the reasons for excluding a subject from an analysis population will be provided on the randomized population by treatment sequence.

The number of subjects reporting at least one major protocol deviation and the number of subjects reporting each considered major PD will be summarized on the randomized


Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

population by treatment sequence and overall. Similarly, the number of subjects reporting at least one minor protocol deviation and the number of subjects reporting each considered minor PD will be summarized on the randomized population by treatment sequence. The list of confirmed protocol deviations and their classification as major/minor was defined in the specific protocol deviation handling plan.



Table 6.1-1:



### **6.2. Background and Demographic Characteristics**

Background and demographic characteristics will be summarized descriptively by treatment sequence and overall on the FAS, mFAS1.





Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021



Medical and surgical history findings will be summarized by System Organ Class and Preferred Term according to the MedDRA dictionary,

Subjects will only be counted once per MedDRA level, and the medical history will be sorted by descending incidence of SOCs and then PTs in the overall group. Medical and surgical history findings will be summarized separately:



In addition, the following variables will be summarized at Visit 1 on the FAS population according to treatment sequence:





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



#### 6.3. Efficacy Evaluation

#### 6.3.1. Primary efficacy analysis

#### **Definition of primary endpoint**

The primary endpoint is the change in weekly global gastrointestinal symptoms average index score from pre-treatment (Baseline/Reference, depending on the period) to the end of each treatment period.

The weekly global gastrointestinal symptoms average index score is obtained by averaging the scores for each of the 4 symptoms assessed weekly: abdominal pain, bloating, nausea and vomiting.

Each symptom (i.e., abdominal pain, bloating, nausea, vomiting) was rated using a recall period of 7 days and a Likert scale with the following categories:

- 0 Absent
- 1 Mild (not influencing usual activities)
- 2 Moderate (diverting from, but not urging modification of, usual activities)
- 3 Severe (influencing usual activities markedly enough to urge modifications)
- 4 Extremely severe (precluding daily activities)





Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

| Considering the evaluable | pairs |
|---------------------------|-------|
| the | |
| will be summarized | |

Of note, each subject should be evaluated twice: once for each cycle. Consequently, each subject can contribute to 0, 1 or 2 pairs and only data that constitute pair evaluable for primary endpoint will be considered in this and in the following analysis.

| Differences | between | velusetrag | and | placebo | will | be | computed | within | each | cycle |
|---|---|---|---|---|---|---|---|---|---|---|

These analyses will be provided on the mFAS1 without any missing data imputation as primary analysis.

Finally, a listing will be provided on Randomized population considering the intake of each collected in the eDiary together with the individual gastrointestinal symptoms and the weekly global gastrointestinal symptoms average index score.

#### Data handling rules

Missing data will be handled as described in Section 4.4.2.

Sensitivity analysis



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



# 6.3.2. Secondary efficacy analysis





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

These analyses will be performed only on mFAS1 and without missing imputation.

#### <u>Definition</u>

The as described in section 6.3.1. will be computed

The proportion of subjects with change between the end of treatment and pretreatment value  $\leq$  - 1 point will be computed and considered as "Success" while the proportion of subjects with change between the end of treatment and pre-treatment value>-1 will be considered as "Failure".

#### Data handling rules

No missing imputation will be performed.

#### **Definition**

Each symptom (i.e., property of the symptom of 7 days and a Likert scale with the following categories:

0 - Absent

1 - Mild (not influencing usual activities)



Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

- 2 Moderate (diverting from, but not urging modification of usual activities)
- 3 Severe (influencing usual activities markedly enough to urge modifications)
- 4 Extremely severe (precluding daily activities)

The endpoint is the score from pre-treatment to the end of each treatment period. A represents improvement. **Definition** The number of and will be provided in the eDiary every 7 days together with the evaluation of the on average according to scale. Changes in the number of and number of will be computed between the end of each treatment period and the pre-treatment (Baseline/Reference).





#### Data handling rules



Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

#### **Definition**

The will be provided in the eDiary every 7 days according to a scale from 0=very unhappy to 10=very happy.

Changes in will be computed between the end of treatment number and the pre-treatment number (Baseline/Reference). A positive change represents an improvement.

#### **Definition**

The will be computed based on the to assess consists in timed and standardized measurement of a solution of water and

This evaluation will be performed only during the first treatment period of the study.

Changes in will be computed between the post-treatment (i.e., end of first treatment period at Visit 3 (EOT-1)) and the pre-treatment (i.e., Screening value at Visit 1).

#### Data handling rules



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

**Definition** levels are . Their levels will be collected at pre-treatment (Baseline/Reference) and at the end of follow-up after the fourth period and at ETV and ESV. Changes in will be computed between the end of each 2week wash-out period (or follow up period) and the relevant pre-treatment values (Baseline/Reference)(i.e., for period 1: levels at V4 – levels at V1; for period 2: levels at V6 – levels at V4; for period 3: levels at V8 – levels at V6 and for period 4: levels at V10 - levels at V8).

### Data handling rules



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### **Definition**

For each intakes: , the subject provides daily the status of the

- Not taken
- Taken at the prescribed dose
- Taken at reduced dose
- Taken at increased dose

the following flag are calculated:

Increase flag: for each day, a drug will be considered as taken at increase dose

Baseline/Reference is defined as the last information collected in the eDiary in the previous phase. It will be Day -1 for Treatment Period 1, the last day in Treatment Period 1 for Wash-out Period 1 and so on.

These flags will be reviewed and updated by means of Medical Review to evaluate if the computed flags are clinically consistent.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



The numerator will be considered as follows:

- Proportion of days with dose increased (at least 1 medication):
- Proportion of days with dose increased (1-2 medications):
- Proportion of days with dose increased (>=3 medications):
- Proportion of days with dose decreased (at least 1 medication):
- Proportion of days with dose decreased (1-2 medications):
- Proportion of days with dose decreased (>=3 medications):
- Proportion of days with drug added (at least 1 medication):
- Proportion of days with drug removed (at least 1 medication):

#### Analysis methodology





Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021

#### Data handling rules

No missing imputation will be performed.

# Definition The used to assess generic outcomes from the subject's perspective. It is often used as a measure. Generic subject-reported outcome (PRO) measures like the including the impact of any and all illnesses on a broad range of functional domains. The consists of a subset of from the covering the same domains of , including (norm based score) that represents will be derived by means of the components of and Analysis methodology

### Data handling rules

No missing imputation will be performed.

# 6.3.2.11.

#### **Definition**

The number of during each treatment period will be collected and analyzed as well as the number of each wash-out/follow-up period.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

#### Analysis methodology



### Data handling rules

No missing imputation will be performed.



### Analysis methodology





Sponsor: Alfasigma S.p.A. Protocol: VE-CIP2001/2021



#### Data handling rules

No missing imputation will be performed.

#### **Definition**

The number of during each treatment period will be collected and analyzed as well as the number of each wash-out/follow-up period.

#### Analysis methodology



#### Data handling rules

No missing imputation will be performed.

<u>Definition</u>

The effect of will be evaluated considering the following set of variables previously described:



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



#### Analysis methodology



#### 6.3.2.15. Concentration of velusetrag and THRX-830449 metabolite

#### **Definition**

Serial blood samples for assessment of will be collected

For each sample, the possible results will be a number indicating the concentration in pg/mL or one of the following other cases: NQ = < Assay LLQ, IS = Insufficient Sample, NR = Not Reportable, or NA =Not Analysed. If results is equal to IS = Insufficient Sample, NR = Not Reportable, NA =Not Analysed or NQ =< Assay LLQ the concentration is not available and will be missing for the summary table and graph.

#### Analysis methodology



#### Data handling rules



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

### **6.3.3.** Exploratory efficacy analysis

Not applicable.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



#### 6.4. Safety Evaluation

The safety analyses will be performed on subjects included in the SS.

#### 6.4.1. Extent of Exposure

Exposure time will be computed in weeks within each period of treatment as follows:

(Last intake date in the study period - First intake date in the study period +1)/7

#### 6.4.2. Concomitant medications

are defined as therapies ending or ongoing after the start of study treatment (i.e., first intake of treatment in the period 1).

will be presented by ATC Code and Preferred Term by actual treatment on the SS, presenting the number and percentage of subjects with at least one concomitant medication.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



Similarly, medications for CIPO will be presented by ATC Code and Preferred Term by actual treatment on the Safety Population, presenting the number and percentage of subjects with at least one medication for CIPO. Subjects will be counted once in each category, outputs will be sorted in the overall group by descending frequencies of ATC and Preferred Term.

#### Non-drug therapies or surgical and medical procedures

Similarly, non-drug therapies or surgical and medical procedures will be summarized by SOC and Preferred Term by actual treatment on the Safety Population,

#### 6.4.3. Adverse Events

Treatment-emergent adverse events (TEAEs) will be reported by actual treatment. Adverse events starting on or after the first intake of treatment (i.e., first intake in the period 1) are considered TEAEs.

the period 1) are considered TEAEs.



Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



In addition, TEAEs will be summarized by actual treatment, MedDRA System Organ Class and Preferred Terms considering:



Adverse events will be classified as velusetrag emergent if the last treatment taken before the start of the adverse event was velusetrag, or placebo emergent if the last treatment taken before the start of the adverse event was placebo.

In addition, a summary of TEAEs will be provided by treatment sequence.

#### 6.4.4. Laboratory parameters

The safety laboratory tests include . The following variables are measured during the study:



Sponsor: Alfasigma S.p.A.
Protocol: VE-CIP2001/2021



Of note, will be collected with different unit of measurements (i.e., sec or ratio). Since there is no conversion factor applicable to uniform the units, these parameters will be summarized separately according to unit of measurements.





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021



#### 6.4.5. Vital signs/Physical examination



#### 6.4.6. Other safety parameters

(e.g., without artifacts) will be performed and the average of the three readings will be used to determine will be reviewed at the clinical center and final interpretation of all will be completed by a central reviewer and sent to the site for Investigators' subject evaluation and filing. This final investigation will be considered for the following analyses:





Sponsor: Alfasigma S.p.A.

Protocol: VE-CIP2001/2021

Pregnancy test and COVID-19 rapid swab will be only listed.

### 6.5. Subgroup Analyses

Not applicable.

### 6.6. Interim Analysis and Data Monitoring

Not applicable.

#### 7. REFERENCES

Not applicable.

#### 8. APPENDIX

Not applicable.

# **DocuSign**

#### **Certificate Of Completion**

Envelope Id: 16D69DD0BF734456ADF0523603E96616

Subject: Complete with DocuSign: VE-CIP2001\_2021\_Statistical\_Analysis\_Plan\_final2.0\_20230510.pdf

Source Envelope:

Document Pages: 59 Certificate Pages: 5

Signatures: 4 Initials: 0

AutoNav: Enabled

**Envelopeld Stamping: Enabled** 

Time Zone: (UTC+01:00) Amsterdam, Berlin, Bern, Rome, Stockholm, Vienna

**Envelope Originator:** 

Status: Completed



IP Address:

#### **Record Tracking**

Status: Original

10-May-2023 | 18:38

Holder:

Location: DocuSign

#### Signer Events

Security Level: Email, Account Authentication

(Required)

Signature

DocuSigned by:

D Signer Name: Signing Reason: I am the author of this document Signing Time: 10-May-2023 | 18:41 CEST **Timestamp** 

Sent: 10-May-2023 | 18:40 Viewed: 10-May-2023 | 18:40 Signed: 10-May-2023 | 18:41

Signature Adoption: Pre-selected Style Signature ID:

Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I am the author of this document

Electronic Record and Signature Disclosure:

Accepted: 10-May-2023 | 18:40

Security Level: Email, Account Authentication (Required)

DocuSigned by:

Signer Name: Signing Reason: I have reviewed this document Signing Time: 10-May-2023 | 18:46 CEST

Sent: 10-May-2023 | 18:41 Viewed: 10-May-2023 | 18:46 Signed: 10-May-2023 | 18:47

Signature Adoption: Pre-selected Style Signature ID:

Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I have reviewed this document

Electronic Record and Signature Disclosure: Accepted: 10-May-2023 | 18:46

Signer Events **Signature** Timestamp Sent: 10-May-2023 | 18:47 Viewed: 10-May-2023 | 19:30 Security Level: Email, Account Authentication Signed: 10-May-2023 | 19:31 (Required) Signature Adoption: Pre-selected Style Signature ID: Using IP Address: With Signing Authentication via DocuSign password With Signing Reasons (on each tab): I approve this document Electronic Record and Signature Disclosure: Accepted: 10-May-2023 | 19:30 ID: Sent: 10-May-2023 | 19:31 Viewed: 10-May-2023 | 22:59 Security Level: Email, Account Authentication Signed: 10-May-2023 | 23:00 (Required)

Signature Adoption: Pre-selected Style Signature ID:

Using IP Address:

With Signing Authentication via DocuSign password With Signing Reasons (on each tab):

I approve this document

Electronic Record and Signature Disclosure: Accepted: 10-May-2023 | 22:59

In Person Signer Events Signature **Timestamp Editor Delivery Events Status** Timestamp **Agent Delivery Events Status Timestamp Intermediary Delivery Events Status** Timestamp **Certified Delivery Events Status Timestamp Carbon Copy Events Status** Timestamp Witness Events Signature **Timestamp Notary Events** Signature **Timestamp Envelope Summary Events Status** Timestamps **Envelope Sent** Hashed/Encrypted 10-May-2023 | 18:40 Certified Delivered Security Checked 10-May-2023 | 22:59 Signing Complete Security Checked 10-May-2023 | 23:00 Completed Security Checked 10-May-2023 | 23:00 **Payment Events Timestamps Electronic Record and Signature Disclosure** 

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through the DocuSign system. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to this Electronic Record and Signature Disclosure (ERSD), please confirm your agreement by selecting the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

#### Getting paper copies

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. You will have the ability to download and print documents we send to you through the DocuSign system during and immediately after the signing session and, if you elect to create a DocuSign account, you may access the documents for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

#### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. Further, you will no longer be able to use the DocuSign system to receive required notices and consents electronically from us or to sign electronically documents from us.

All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through the DocuSign system all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

### How to contact:

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to:

### To advise of your new email address

To let us know of a change in your email address where we should send notices and disclosures electronically to you, you must send an email message to us at and in the body of such request you must state: your previous email address, your new email address. We do not require any other information from you to change your email address.

If you created a DocuSign account, you may update it with your new email address through your account preferences.

# To request paper copies from

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an email to and in the body of such request you must state your email address, full name, mailing address, and telephone number. We will bill you for any fees at that time, if any.

# To withdraw your consent with

To inform us that you no longer wish to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your signing session, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may;

ii. send us an email to and in the body of such request you must state your email, full name, mailing address, and telephone number. We do not need any other information from you to withdraw consent. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

The minimum system requirements for using the DocuSign system may change over time. The current system requirements are found here: <a href="https://support.docusign.com/guides/signer-guide-signing-system-requirements">https://support.docusign.com/guides/signer-guide-signing-system-requirements</a>.

#### Acknowledging your access and consent to receive and sign documents electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please confirm that you have read this ERSD, and (i) that you are able to print on paper or electronically save this ERSD for your future reference and access; or (ii) that you are able to email this ERSD to an email address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format as described herein, then select the check-box next to 'I agree to use electronic records and signatures' before clicking 'CONTINUE' within the DocuSign system.

By selecting the check-box next to 'I agree to use electronic records and signatures', you confirm that:

- You can access and read this Electronic Record and Signature Disclosure; and
- You can print on paper this Electronic Record and Signature Disclosure, or save or send this Electronic Record and Disclosure to a location where you can print it, for future reference and access; and
- Until or unless you notify as described above, you consent to receive exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you by during the course of your relationship with